CLINICAL TRIAL: NCT00518349
Title: Evaluation of a Novel Colonoscope Designed for Easier Passage Through Flexures: A Randomised Study
Brief Title: Colonoscope Passive Bending Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Department of Health and Social Affairs (Other Government)
Collaborators: Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Geir Hoff, Head of Research, Telemark Hospital, Norwegian Department of Health and Social Affairs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ST161006
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Results first posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2017-09

CONDITIONS: Colitis; Adenoma; Carcinoma; Functional Colonic Disease
MeSH Terms: conditions — Colitis; Adenoma; Carcinoma; Colonic Diseases, Functional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prototype colonoscope (Active Comparator): Colonoscopy using prototype colonoscope with passive bending function
  Interventions: Device: Passive bending function
- Standard colonoscope (Placebo Comparator): Colonoscopy using standard colonoscope with no passive bending function
  Interventions: Device: No passive bending function

INTERVENTIONS:
Device: Passive bending function — Colonoscope with a passive bending function
  Other Names: passive bending colonoscope
  Arms: Prototype colonoscope
Device: No passive bending function — Examination using standard colonoscope without passive bending function
  Other Names: standard colonoscope
  Arms: Standard colonoscope

SUMMARY:
A prototype colonoscope with an extra passively bending distal section has been developed by Olympus Japan (ref. publications). The present study (2006-2007) is testing refinements of this function.

DETAILED DESCRIPTION:
Results from the first prototype evaluation has been published.Modifications are presently evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for routine outpatients colonoscopy

Exclusion Criteria:

* Pregnant women
* Age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-08; Primary Completion 2007-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geir Hoff, MD, PhD, Principal Investigator — Head of Research, Telemark Hospital
Locations (1):
- Gastroenterology section, Dept. of Medicine, Telemark Hospital, Skien, Norway

REFERENCES:
- [Background] Hoff G, Moritz V, Bretthauer M, Ludolph T, Huppertz-Hauss G, Paulsen J, Seip B, Sauar J, Kjellevold O, Chengarov L. Colonoscope with a sub-distal hyper-flaccid segment for improved insertion at colonoscopy: a randomized study. Scand J Gastroenterol. 2011 Jan;46(1):104-8. doi: 10.3109/00365521.2010.521891. Epub 2010 Oct 6. PMID 20923378
- [Result] Hoff G, Bretthauer M, Huppertz-Hauss G, Sauar J, Paulsen J, Dahler S, Kjellevold O. Evaluation of a novel colonoscope designed for easier passage through flexures: a randomized study. Endoscopy. 2005 Nov;37(11):1123-6. doi: 10.1055/s-2005-870444. PMID 16281143

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 120 patients, routinely referred for outpatients colonosciopy, were randomized 1:1 to examination with protototype or standard colonoscope.
Pre-assignment Details: Exclusion criteria were pregnancy, age younger than 18 years, previous resection for colorectal disease and inability to comprehend the information given.
Groups:
- Prototype Colonoscope: Colonoscopy using prototype colonoscope
- Standard Colonoscope: Colonoscopy using standard colonoscope without a passive bending function
Period: Overall Study
Arm/Group | Prototype Colonoscope | Standard Colonoscope
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients referred to routine outpatients' colonoscopy
Groups:
- 1 Prototype Colonoscope: Colonoscopy using prototype colonoscope
- 2 Standard Colonoscope: Colonoscopy using standard colonoscope without a passive bending function
- Total: Total of all reporting groups
Arm/Group | 1 Prototype Colonoscope | 2 Standard Colonoscope | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 35 | 73
  >=65 years | 22 | 25 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (15.4) | 58.6 (17.6) | 58.8 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 31 | 30 | 61
Region of Enrollment [Number; unit: participants]
  Norway | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Patient Assessment of Pain Experienced During Colonoscopy
Description: The proportion of patients reporting "no pain" when examined with prototype or standard colonoscope, respectively. Pain experienced was assessed by the patient in a questionnaire to be filled in at home on the day after the examination and mailed in a pre-paid envelope to a national quality register (Gastronet).
Time Frame: Pain experienced during colonoscopy
Population: Power estimates based on assumption of 20% difference in pain-free examination comparing groups
Measure: Number; unit: participants
Arm/Group | 1 Prototype Colonoscope | 2 Standard Colonoscope
Number analyzed (Participants) | 60 | 60
participants | 19 | 10

ADVERSE EVENTS:
Time Frame: Adverse event registration was based on events observed during the patient's stay in the endoscopy unit and information from a patient report form to be filled in by the patient on the day after the examination.
Description: Patients were provided with a patient report form to be returned to the national quality assurance register Gastronet in a prepaid return envelope on the day after the colonoscopy.
Groups:
- Prototype Colonoscope: The prototype colonoscope is in effect a standard Olympus endoscope with one exception: about 10cm proximal to the distal, actively bending tip, there is a more falccid section which bends passively in all directions against external pressure. It is hypothesized that this will ease passage through sharp bends (flexures).
- Standard Colonoscope: Colonoscope without a distal actively bending section
Arm/Group | Prototype Colonoscope | Standard Colonoscope
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No